CLINICAL TRIAL: NCT03987308
Title: Comparing the Efficacy and Safety Between Short-term Continuous Subcutaneous Beinaglutide Injection and Continuous Subcutaneous Insulin Infusion (CSII) for Treatment of Patients With Newly Diagnosed Type 2 Diabetes: a Multicenter, Randomized Open Trial Study With Parallel Controls
Brief Title: Comparing the Efficacy and Safety Between Continuous Subcutaneous Beinaglutide and CSII for Newly Diagnosed T2DM Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BN-IIT-IS-008
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetic Patients; T2DM (Type 2 Diabetes Mellitus); T2DM
Keywords: T2DM; beinaglutide; CSII; subcutaneous pump
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glucagon-like peptide 1 (7-36); Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Beinaglutide infusion (Experimental): 8-week Beinaglutide (continuous subcutaneous infusion) treatment group
  Interventions: Drug: Beinaglutide
- Continuouns Insulin aspart infusion (Active Comparator): 8-week insulin aspart (CSII) treatment group
  Interventions: Drug: Insulin aspart

INTERVENTIONS:
Drug: Beinaglutide — Beinaglutide (continuous subcutaneous infusion)
  Arms: Continuous Beinaglutide infusion
Drug: Insulin aspart — Insulin aspart (CSII)
  Arms: Continuouns Insulin aspart infusion

SUMMARY:
The efficacy, safety and post-treatment disease control will be compared between groups of continuous subcutaneous Beinaglutide infusion and continuous subcutaneous insulin infusion (CSII) in adult patients with newly diagnosed type 2 diabetes.

DETAILED DESCRIPTION:
Based on the dual roles of glucagon-like peptide 1 (GLP-1) in regulating fasting blood glucose and postprandial blood glucose secretion, we adopted a combinational therapeutic model and will administer drug treatments during meals. Newly diagnosed type 2 diabetic patients will be administered continuous subcutaneous Beinaglutide injections using a pump device. The efficacy, safety and disease control after terminating the drug treatments will be compared to those of patients who receive CSII treatment.

This is a national-level, multicenter, randomized, open study with parallel controls. The study consists of two phases:

a 8-week treatment phase and a 12-week post-treatment follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years (inclusive) at enrollment, regardless of gender.
2. Voluntary signing of the informed consent form.
3. Newly diagnosed type 2 diabetes mellitus patients, diagnosed according to the WHO 1999 criteria, with a disease duration ≤1 year.
4. HbA1c between 7.5% and 10.0%.
5. BMI between 24 kg/m² and 42 kg/m².
6. Subjects who have not taken antidiabetic medications or have used oral antidiabetic medications for less than 3 months and have discontinued for more than 1 month (calculated from the date of signing the informed consent form).
7. Subjects with reproductive potential (including male subjects whose partners have reproductive potential) agree to use effective contraception during the study and for 1 month after study completion.

Exclusion Criteria:

1. Patients with type 1 diabetes or other types of diabetes.
2. History of obstructive intestinal diseases or potential complications: subjects with post-abdominal surgery or peritoneal infection-related intestinal adhesions, intestinal obstruction sequelae; subjects with intestinal motility disorders, chronic constipation; subjects with a history of Crohn's disease or ulcerative colitis.
3. History of pancreatitis.
4. Family history of medullary thyroid carcinoma.
5. History of malignant tumors.
6. ALT, AST >3 times the upper limit of normal, and/or total bilirubin >2 times the upper limit of normal.
7. Moderate to severe renal insufficiency (eGFR <60 ml/min/1.73m²).
8. Triglycerides ≥5.0 mmol/L.
9. Multiple endocrine neoplasia type 2 (MEN 2).
10. Participation in any pre-marketing drug study within 3 months.
11. Use or expected use of systemic corticosteroids, immunosuppressants, or cytotoxic drugs during the study period.
12. History of diabetic ketoacidosis or non-ketotic hyperosmolar coma within 6 months prior to screening.
13. Blood pressure exceeding the following criteria (untreated or treated): systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg.
14. History of any of the following cardiovascular diseases within 3 months prior to screening: acute myocardial infarction, New York Heart Association functional class III/IV heart failure or left ventricular ejection fraction ≤40%, or cerebrovascular event (stroke).
15. Allergy to binaclotide or any component of the study drug, or allergy to insulin or any component of the insulin used in the study.
16. Presence of other severe diseases that may interfere with the study, as judged by the investigator.
17. Pregnant or breastfeeding women.
18. Poor compliance, as judged by the investigator, and inability to complete the study as required.
19. Inability to undergo continuous pump infusion: subjects allergic to subcutaneous infusion tubes or adhesive tape; subjects unwilling to have long-term subcutaneous infusion tubes or continuous pump use; subjects with psychological aversion to pump therapy; subjects or their families lack relevant knowledge and are unable to master the use after training; subjects with severe psychological disorders or mental abnormalities; subjects who are unable to care for themselves and have no caregivers.
20. Any other factors deemed unsuitable for participation in the study by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2019-07-02 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects achieving HbA1c <7.0%, no weight increase (≤0 kg), and no hypoglycemia (blood glucose ≤3.9 mmol/L or severe hypoglycemia) after 8 weeks of treatment. | From baseline to the end of treatment at 8 week
  The primary endpoint of the trial is a composite endpoint of HbA1c <7.0%, no weight increase (≤0 kg), and no hypoglycemia (blood glucose ≤3.9 mmol/L or severe hypoglycemia) after 8 weeks of treatment..

SECONDARY OUTCOMES:
Proportion of subjects achieving HbA1c reduction <7% after 8 weeks of treatment. | From baseline to the end of treatment at 8 week
  Proportion of participants achieving a reduction in HbA1c levels to below 7% after 8 weeks of treatment.
Changes in fasting blood glucose from baseline after 8 weeks of treatment. | From baseline to the end of treatment at 8 week
  Changes in fasting blood glucose from baseline after 8 weeks of treatment.
Changes in postprandial blood glucose from baseline after 8 weeks of treatment. | From baseline to the end of treatment at 8 week
  Changes in postprandial blood glucose from baseline after 8 weeks of treatment.
Changes in HbA1C from baseline after 8 weeks of treatment. | From baseline to the end of treatment at 8 week
  Changes in HbA1C from baseline after 8 weeks of treatment.
Proportion of subjects with weight reduction ≥5% from baseline after 8 weeks of treatment. | From baseline to the end of treatment at 8 week
  Proportion of subjects with weight reduction ≥5% from baseline after 8 weeks of treatment.
Changes in weight from baseline after 8 weeks of treatment. | From baseline to the end of treatment at 8 week
  Changes in weight from baseline after 8 weeks of treatment.
Changes in waist circumference from baseline after 8 weeks of treatment. | From baseline to the end of treatment at 8 week
  Changes in waist circumference from baseline after 8 weeks of treatment.
Changes in waist-to-hip ratio from baseline after 8 weeks of treatment. | From baseline to the end of treatment at 8 week
  Changes in waist-to-hip ratio from baseline after 8 weeks of treatment.
Changes in fasting insulin from baseline after 8 weeks of treatment. | From baseline to the end of treatment at 8 week
  Changes in fasting insulin from baseline after 8 weeks of treatment.
Changes in fasting C-peptide from baseline after 8 weeks of treatment. | From baseline to the end of treatment at 8 week
  Changes in fasting C-peptide from baseline after 8 weeks of treatment.
Changes in HOMA-β from baseline after 8 weeks of treatment. | From baseline to the end of treatment at 8 week
  Changes in HOMA-β from baseline after 8 weeks of treatment.
Changes in HOMA-IR from baseline after 8 weeks of treatment. | From baseline to the end of treatment at 8 week
  Changes in HOMA-IR from baseline after 8 weeks of treatment.
Changes in lipid profile from baseline after 8 weeks of treatment. | From baseline to the end of treatment at 8 week
  Changes in lipid profile from baseline after 8 weeks of treatment.
Changes in blood pressure baseline after 8 weeks of treatment. | From baseline to the end of treatment at 8 week
  Changes in blood pressure (assessing both of systolic and diastolic pressure) from baseline after 8 weeks of treatment.
Changes in heart rate from baseline after 8 weeks of treatment. | From baseline to the end of treatment at 8 week
  Changes in heart rate from baseline after 8 weeks of treatment.
Proportion of subjects achieving HbA1c <6.5% at 20 weeks. | From baseline to week 20
  Proportion of subjects achieving HbA1c <6.5% at 20 weeks.
Proportion of subjects achieving HbA1c <7% at 20 weeks. | From baseline to week 20
  Proportion of subjects achieving HbA1c <7% at 20 weeks.
Proportion of subjects with fasting blood glucose <7.0 mmol/L at 20 weeks. | From baseline to week 20
  Proportion of subjects with fasting blood glucose <7.0 mmol/L at 20 weeks.
Changes in weight from baseline at 20 weeks. | From baseline to week 20
  Changes in weight from baseline at 20 weeks.
Changes in BMI from baseline at 20 weeks. | From baseline to week 20
  Changes in BMI from baseline at 20 weeks.
Changes in waist-to-hip ratio from baseline at 20 weeks. | From baseline to week 20
  Changes in waist-to-hip ratio from baseline at 20 weeks.
Changes in fasting blood glucose from baseline at 20 weeks. | From baseline to week 20
  Changes in fasting blood glucose HbA1c from baseline at 20 weeks.
Changes in postprandial blood glucose from baseline at 20 weeks. | From baseline to week 20
  Changes in postprandial blood glucose from baseline at 20 weeks.
Changes in HbA1c from baseline at 20 weeks. | From baseline to week 20
  Changes in HbA1c from baseline at 20 weeks.
Changes in HOMA-β from baseline at 20 weeks. | From baseline to week 20
  Changes in HOMA-β from baseline at 20 weeks.
Changes in HOMA-IR from baseline at 20 weeks. | From baseline to week 20
  Changes in HOMA-IR from baseline at 20 weeks.
Changes in fasting insulin from baseline at 20 weeks. | From baseline to week 20
  Changes in fasting insulin from baseline at 20 weeks.
Changes in fasting C-peptide from baseline at 20 weeks. | From baseline to week 20
  Changes in fasting C-peptide from baseline at 20 weeks.
Changes in lipid profile from baseline at 20 weeks. | From baseline to week 20
  Changes in lipid profile from baseline at 20 weeks.

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - Pinggu District Hospital, Beijing, Beijing Municipality
  - Capital Medical University Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - Emergency General Hospital, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - Harbin Medical University Second Hospital, Harbin, Heilongjiang
  - Southeast University Zhongda Hospital, Nanjing, Jiangsu
  - Xuzhou Medical University Affiliated Hospital, Xuzhou, Jiangsu
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - Jilin University Second Hospital, Changchun, Jilin
  - Xi'an Jiaotong University Second Hospital, Xi'an, Shaanxi
  - Southwest Medical University Affiliated Hospital, Luzhou, Sichuan
  - Peking University Binhai Hospital, Tianjin, Tianjin Municipality
  - First Hospital of Peking University, Beijing
  - Heilongjiang provincial hospital, Harbin
  - Henan People's Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No